CLINICAL TRIAL: NCT02340741
Title: Assessing of Carbon Dioxide Insufflation on the Neurological Complications During Open Heart Operations
Brief Title: Insufflation of Carbon Dioxide During Cardiac Surgery as Prevention Neurologic Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11-54-22
Record Dates: First submitted 2014-12-16; First posted 2015-01-19 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Air Embolism; Neurological Damage
Keywords: carbon dioxide; postoperative cerebrovascular complications; air embolism
MeSH Terms: conditions — Embolism, Air; Trauma, Nervous System | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional prophylaxis of aeroembolism (Other): Procedure: cardiac surgery with opening of heart chambers.
  Will be including 167 patients to undergo cardiac surgery. After the main operation phase all heart cavities are sealed, left vent drainage is stopped, ascending aorta is punctured and cardiac massage is performed, ventilation is started and the heart is filled with volume. Operating table is positioned in the Trendelenburg position, and aorta is opened. The amount of air in the cavities is evaluated by transesophageal echocardiography.
  Interventions: Procedure: conventional prophylaxis of aeroembolism; Procedure: cardiac surgery with opening of heart chambers
- conventional prophylaxis plus CO2 insufflation (Other): Procedure: cardiac surgery with opening of heart chambers.
  Will be including 167 patients to undergo cardiac surgery. After the main phase of the operation standard measures of aeroembolism prevention are carried out. The amount of air in the cavities is evaluated by transesophageal echocardiography.
  Interventions: Procedure: conventional prophylaxis plus CO2 insufflation; Procedure: cardiac surgery with opening of heart chambers

INTERVENTIONS:
Procedure: conventional prophylaxis of aeroembolism — 167 patients will be enrolled. Will perform standard way of aeroembolism prevention
  Arms: conventional prophylaxis of aeroembolism
Procedure: conventional prophylaxis plus CO2 insufflation — 167 patients will be enrolled. Will perform standard way of aeroembolism prevention and insufflation of carbon dioxide
  Arms: conventional prophylaxis plus CO2 insufflation
Procedure: cardiac surgery with opening of heart chambers — Patients with different clinical diagnoses, which is planned to cardiac surgery with the opening heart cavities

SUMMARY:
Effect of intraoperative insufflation of carbon dioxide on the neurologic complications in the early postoperative period after open cardiac surgery.

DETAILED DESCRIPTION:
Arterial air embolism in cardiac surgery is not a rare complication, leading to neurological damage in the early postoperative period of 3-5%. Insufflation of carbon dioxide (CO2) into the operative field to prevent cerebral or myocardial damage by air embolism is reported since 1967 in open heart surgery (Selman MW et al. 1967).

Carbon dioxide fills the thoracic cavity by gravity and replaces air if adequately insufflated. Because solubility of CO2 is better than that of air, occlusion or flow disruption in arteries of the brain or the heart is thought to be diminished. Despite carefully performed deairing procedures as puncturing of the ascending aorta and cardiac massage, transcranial Doppler studies revealed large amounts of emboli during the first ejections of the beating heart (van der Linden J et al. 1991). In patiens with minimally invasive approach and redo valve surgery, deairing of the cardiac chambers has become more difficult.

Although the use of carbon dioxide when filling in the surgical field, as the prevention of air embolism reduces the number of intracardiac emboli according to transesophageal echocardiography there is no evidence of a sustained reduction in cerebrovascular events (G. Salvatore al. 2009).

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Informed Consent and Release of Medical Information forms
* Age 18 - 70 years
* Patients scheduled on cardiac surgery with opening cavities

Exclusion Criteria:

* History of stroke and TIA
* Significant carotid artery stenosis
* Presence of initial severe encephalopathy
* Re-clamping of the aorta
* Emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
postoperative neurological disorders (stroke, psychosis,encephalopathy), as measured by Confusion Assessment Method for the ICU, Richmond Agitation-Sedation Scale, Standardized Mini-Mental State Examination | 14 days
  conducting tests: Confusion Assessment Method for the ICU, Richmond Agitation-Sedation Scale, Standardized Mini-Mental State Examination

SECONDARY OUTCOMES:
hospital mortality | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr V Bogachev-Prokophiev, PhD, Principal Investigator — Meshalkin Research Institute of Pathology of Circulation
Locations (1):
- Novosibirsk State Research Institute of Circulation Pathology, Novosibirsk, Novosibirsk Territory, Russia